CLINICAL TRIAL: NCT00003369
Title: Evaluation of Intravenously Administered Tirapazamine Plus Cisplatin in Cervical Cancer
Brief Title: S9717 Tirapazamine Plus Cisplatin in Treating Patients With Metastatic, Recurrent, or Refractory Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066358; SWOG-S9717 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-06-24 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Cervical Cancer
Keywords: stage IV cervical cancer; recurrent cervical cancer; cervical squamous cell carcinoma; cervical adenosquamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Tirapazamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tirapazamine/cisplatin (Experimental): tirapazamine and cisplatin given Day 1 of each 21-day treatment cycle
  Interventions: Drug: cisplatin; Drug: tirapazamine

INTERVENTIONS:
Drug: cisplatin — 75 mg/m2 IV as a one-hour infusion after tirapazamine on Day 1 of each 21-day cycle
  Other Names: platinol
Drug: tirapazamine — 260 mg/m2 over two hours prior to cisplatin on Day 1 of each 21-day cycle

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy consisting of tirapazamine plus cisplatin in treating patients who have metastatic, recurrent, or refractory cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the survival of patients with metastatic or recurrent epithelial squamous or adenosquamous carcinoma of the cervix when treated with intravenous tirapazamine plus intravenous cisplatin. II. Evaluate the unconfirmed complete and partial response rates of these patients, as well as, the nature and degree of toxicity associated with this regimen in this patient population.

OUTLINE: Patients receive tirapazamine intravenously over 2 hours and then, following a 1 hour rest, receive cisplatin intravenously over 1 hour. Courses are repeated every 21 days. Treatment continues for 6-10 courses in the absence of unacceptable toxic effects or disease progression. All patients are followed every 6 months for 2 years, then annually thereafter until death.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed squamous or adenosquamous carcinoma of the cervix that is metastatic, recurrent, or refractory Any stage disease treated with prior radical surgery and/or definitive radiotherapy that has locally recurred and is no longer amenable to surgery or radiotherapy OR Metastatic disease that is not amenable to surgery or radiation therapy Measurable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Not specified Renal: Creatinine no greater than 1.5 times upper limit of normal Other: No history of allergic reaction to mannitol Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 3 months after study No other prior malignancy except: Adequately treated basal cell or squamous cell skin cancer In situ cervical cancer Adequately treated stage I or II cancer from which the patient is currently in complete remission Any other cancer from which the patient has been disease free for 5 years

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent colony stimulating factor therapy Chemotherapy: Prior chemotherapy (hydroxyurea, fluorouracil, metronidazole, cisplatin, or other platinum agent) allowed as a radiosensitizing agent only No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Prior radiotherapy allowed to less than 30% of the bone marrow only Recovered from toxic effects No concurrent radiotherapy Surgery: See Disease Characteristics Prior surgery allowed Recovered from effects of prior surgery Other: No prior systemic therapy for this disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 1998-08; Primary Completion 2003-10 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
overall survival | 6 months
  From date of registration to date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Harriet O. Smith, MD, Study Chair — University of New Mexico Cancer Center
Locations (85):
- United States (85):
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Smith HO, Jiang CS, Weiss GR, Hallum AV 3rd, Liu PY, Robinson WR 3rd, Cheng PC, Scudder SA, Markman M, Alberts DS. Tirapazamine plus cisplatin in advanced or recurrent carcinoma of the uterine cervix: a Southwest Oncology Group study. Int J Gynecol Cancer. 2006 Jan-Feb;16(1):298-305. doi: 10.1111/j.1525-1438.2006.00339.x. PMID 16445649
- [Result] Smith HO, Jiang C, Weiss GR, et al.: Tirapazamine plus cisplatin in advanced or recurrent squamous or adenosquamous carcinoma of the uterine cervix: a phase II study of the Southwest Oncology Group. [Abstract] Gynecol Oncol 92 (1): A-49, 416, 2004.